CLINICAL TRIAL: NCT05569603
Title: Effects of Chronobiology-guided Lifestyle Interventions on Insomnia Severity, Cognitive Performance, and Sleepiness in Female Rotating-shift Nurses: a Randomized Controlled Trial
Brief Title: Effects of Chronobiology-guided Lifestyle Interventions on Insomnia Severity, Cognitive Performance, and Sleepiness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: Taipei Medical University (Other); Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2021-06-002A
Record Dates: First submitted 2021-09-06; First posted 2022-10-06 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Circadian Rhythm Sleep Disorder
Keywords: Chonobiology; Cognitive performance; Insomnia; Shift work; Sleepiness
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm; Sleep Initiation and Maintenance Disorders; Sleepiness

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chronobiology-guided lifestyle interventions group (Experimental): A multimodal program that includes (1) timed bright light therapy, (2)guidance on meal timing, and (3) sleep hygiene education.
  Interventions: Behavioral: Chronobiology-guided lifestyle interventions
- wait-list control group (No Intervention): The participants in the wait-list group will be told that they are on a waiting list during the first 2 weeks to serve as the no-treatment control. Chronobiology-guided lifestyle interventions will be conducted after the posttest is completed.

INTERVENTIONS:
Behavioral: Chronobiology-guided lifestyle interventions — 1) timed bright light exposure using blue-enriched white light glasses, 2) recommendations for meal timing, and 3) sleep hygiene education
  Arms: Chronobiology-guided lifestyle interventions group

SUMMARY:
Poor sleep is closely related to circadian misalignment; shift workers often experience shift work disorder characterized by excessive sleepiness and recurrent shift work schedules-associated insomnia. This study aims to examine the effects of a program of chronobiology-guided lifestyle interventions (CGLI) on insomnia severity, cognitive performance (psychomotor vigilance and processing speed), and sleepiness in female nurses undertaking rotating-shift work.

DETAILED DESCRIPTION:
This study will use a parallel-group, randomized, assessor-blind, wait-list controlled design to determine the effects of a program of multimodal lifestyle interventions based on chronobiology, consisting of timed bright light exposure, meal timing manipulations, and sleep hygiene education on insomnia severity, cognitive performance (psychomotor vigilance and processing speed), and sleepiness in female nurses undertaking rotating-shift work.

ELIGIBILITY:
Inclusion Criteria:

1. Females aged 20 to 60 who work full time as a nurse and work a 3-shift rotation, including day shifts, evening shifts, and night shifts in the most recent 6 months.
2. Participants must complain of insomnia symptoms and/or sleepiness in relation to shift work schedule for at least 3 months.
3. Participants must have10 workdays (evening or night shift) within a 14-day period during the study period.

Exclusion Criteria:

1. Active physical diseases.
2. Moderate to severe psychopathology.
3. Medications or treatments that may affect sleep.
4. Pregnant or breastfeeding.
5. Participants must be free of ophthalmic pathology, eye surgery, and diseases affecting the retina or taking photosensitizing drugs.
6. Participants who have been diagnosed with sleep-disordered breathing will be excluded. Sleep-disordered breathing such as obstructive sleep apnea (OSA) will be screened using the snoring, tiredness, observed apnea, high BP, BMI, age, neck circumference, and male gender (STOP-BANG) questionnaire.

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 80 (Estimated)
Dates: Start 2022-01-12 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
insomnia severity | Through study completion, an average of 14days
  The Insomnia Severity Index will be used to determine the severity of insomnia. The Insomnia Severity Index with a total score ranging from 0 to 28. A higher Insomnia Severity Index score indicates more severe insomnia.

SECONDARY OUTCOMES:
The neurobehavioral function of cognitive performance | Through study completion, an average of 14 days
  The neurobehavioral function will be evaluated using the Walter Reed Psychomotor Vigilance Test (PVT), a portable reaction-time test based on the Dinges and Powell digital test. The PVT will be testing a 5-min test with responses to randomly spaced stimuli per test.
The processing speed of cognitive performance | Through study completion, an average of 14 days
  A Tablet-based Symbol Digit Modalities Test (T-SDMT) will be used to test processing speed.
The sleepiness at work | Through study completion, an average of 14 days
  The Karolinska Sleepiness Scale (KSS) will be used to measure sleepiness at work. It is on a scale of 1 to 9. A higher score is more sleepy.

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Shan Tsai, Professor, Study Chair — Taipei Medical University; Shan-Ying Wu, Master, Principal Investigator — Taipei Vetern General Hospital
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No